CLINICAL TRIAL: NCT00676585
Title: Corticosteroids Therapy in Refractory Shock Following Cardiac Arrest
Brief Title: Corticosteroid Therapy in Refractory Shock Following Cardiac Arrest
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michael Donnino, Michael Donnino, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007P000227
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest, Shock, Steroids
MeSH Terms: conditions — Heart Arrest; Shock | interventions — Saline Solution; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Normal Saline
  Interventions: Drug: Normal Saline
- 1 (Experimental): Hydrocortisone 100mg every 8 hours.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Normal Saline — Normal Saline
  Arms: 2
Drug: Hydrocortisone — Hydrocortisone 100mg
  Arms: 1

SUMMARY:
The major goal of this project is to determine whether the use of physiologic doses of corticosteroids will decrease time to shock reversal, alters the inflammatory cascade, and alters microcirculatory flow in post-cardiac arrest patients.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Either pre-hospital cardiac arrest and ROSC or Inpatient Cardiac Arrest with resultant ROSC
* Vasopressor dependent for a minimum of 1 hour post-arrest

Exclusion Criteria:

* Pregnant
* Indication for Corticosteroids outside of current research proposal
* DNR or comfort care measures
* Presence of septic shock
* Chronic Use (>1week) of oral Corticosteroids in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Donnino MW, Andersen LW, Berg KM, Chase M, Sherwin R, Smithline H, Carney E, Ngo L, Patel PV, Liu X, Cutlip D, Zimetbaum P, Cocchi MN; Collaborating Authors from the Beth Israel Deaconess Medical Center's Center for Resuscitation Science Research Group. Corticosteroid therapy in refractory shock following cardiac arrest: a randomized, double-blind, placebo-controlled, trial. Crit Care. 2016 Apr 3;20:82. doi: 10.1186/s13054-016-1257-x. PMID 27038920

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Normal Saline
- Intervention: Hydrocortisone
Period: Overall Study
Arm/Group | Control | Intervention
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (13) | 66 (15) | 69 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time to Shock Reversal
Description: The primary outcome was time to shock reversal defined as at least 24 hours off all vasopressor medications.
Time Frame: 7 Days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
hours | 55 [30 to 59] | 49 [25 to 71]

2. Secondary Outcome: Mortality
Time Frame: Length of hospital stay, an average of 9 days with a maximum of 36 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
Participants | 16 | 18

3. Secondary Outcome: Sub-group Analysis of Patients With Adrenal Insufficiency
Description: Sub-analysis of patients with adrenal insufficiency: absolute insufficiency as defined by a baseline cortisol level < 15 ug/dL
Time Frame: At time of enrollment
Population: There were 9 patients identified with baseline absolute cortisol deficiency (3 in the control arm and 6 in the intervention arm). This sub population of study participants were analyzed for shock reversal, good neurological outcomes, and survival as shown in each row of the table below.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 3 | 6
Participants
  Shock Reversal in Adrenal Insufficient | 1 | 6
  Good Neurological Outcome in Adrenal Insufficient | 0 | 2
  Survival in Adrenal Insufficient | 0 | 3

ADVERSE EVENTS:
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 16/25 | 18/25
Other Adverse Events (participants affected / at risk) | 19/25 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=25) | Intervention (N=25)
Death (General disorders) | 16 | 18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=25) | Intervention (N=25)
New or Changed Antibiotics (Infections and infestations) | 11 | 9
New insulin infusion (Endocrine disorders) | 6 | 7
Any Bleeding (General disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes